CLINICAL TRIAL: NCT05713058
Title: Effects of Early Time-restricted Carbohydrate Consumption on Weight Loss and Glucose Homeostasis in Patients With Type 2 Diabetes
Brief Title: Metabolic Effects of Early Time-restricted Carbohydrate Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Andrea Natali, Full Professor of Nutrition, Azienda Ospedaliero, Universitaria Pisana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: eTRC DIET
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Diabetes Mellitus, Type 2; Obesity; Nutrition, Healthy; Weight Loss
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eTRC diet (Experimental)
  Interventions: Behavioral: eTRC diet
- Control diet (Active Comparator)
  Interventions: Behavioral: Control diet

INTERVENTIONS:
Behavioral: eTRC diet — 12-week dietary prescription with moderate energy restriction (approximately 200 kcal/day) focusing on the distribution of macronutrients within the day so as to avoid carbohydrate consumption after lunch
  Arms: eTRC diet
Behavioral: Control diet — 12-week dietary prescription with moderate energy restriction (approximately 200 kcal/day) without any recommendations on the distribution of macronutrients within the day
  Arms: Control diet

SUMMARY:
In this clinical trial, the investigators aim to examine the impact of a 12-week early time-restricted carbohydrate consumption diet on weight loss and glucose metabolism in patients with overweight/obesity and type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* age 18-75 years
* both males and females
* type 2 diabetes

Exclusion Criteria:

* type 1 diabetes
* insulin treatment
* pharmacological treatment for weight loss
* pregnancy
* other acute or chronic conditions influencing body weight and glucose metabolism

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Glycemic control | 12 weeks
  Change in plasma levels of glycated hemoglobin

SECONDARY OUTCOMES:
Glucose tolerance | 12 weeks
  Glucose tolerance will be measured as the area under the curve of plasma glucose levels in response to a 180-minute mixed meal tolerance test (MMTT)
Body weight loss | 12 weeks
  Change in body weight

OTHER OUTCOMES:
Daily glucose variability | 14 days
  Glucose variability will be measured as the coefficient of variation (CV) of glucose levels recorded by continuous glucose monitoring over a 14-day period using a FreeStyle Libre 2 sensor
Beta cell function | 12 weeks
  Beta cell function will be measured as the beta cell glucose sensitivity obtained from mathematical modeling of plasma glucose and C-peptide levels in response to a 180-minute mixed meal tolerance test (MMTT)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natali, MD, Principal Investigator — University of Pisa
Locations (1):
- Azienda Ospedaliero-Universitaria Pisana, Pisa, PI, Italy

IPD SHARING:
Plan to Share IPD: No
IPD will be shared with other researchers only upon reasonable request to the PI

REFERENCES:
- [Derived] Trico D, Masoni MC, Baldi S, Cimbalo N, Sacchetta L, Scozzaro MT, Nesti G, Mengozzi A, Nesti L, Chiriaco M, Natali A. Early time-restricted carbohydrate consumption vs conventional dieting in type 2 diabetes: a randomised controlled trial. Diabetologia. 2024 Feb;67(2):263-274. doi: 10.1007/s00125-023-06045-9. Epub 2023 Nov 16. PMID 37971503